CLINICAL TRIAL: NCT03822494
Title: CyberKnife Dose Escalation for Unfavorable and High-risk Prostate Cancer
Brief Title: CyberKnife Dose Escalation Prostate Cancer Trial
Acronym: CK-DESPOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Crozer-Keystone Health System (Other)
Responsible Party: Principal Investigator, Rachelle Lanciano M.D., Principal Investigator, Crozer-Keystone Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCK-02
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Neoplasm
Keywords: radiation therapy; Cyberknife; SBRT; Protons
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dose Escalated CyberKnife SBRT (Experimental): DE-SBRT will be delivered using the CyberKnife robotic radiosurgery system. Patients will be treated with five SBRT treatments (8 Gy per fraction to the PTV, and 9-10 Gy per fraction to any nodules identified on endorectal MRI) over 7-10 days.
  Interventions: Radiation: CyberKnife SBRT

INTERVENTIONS:
Radiation: CyberKnife SBRT — Radiation Therapy

SUMMARY:
Stereotactic body radiation therapy (SBRT) has been employed in the treatment of prostate cancer. Multiple single institution experiences suggest high biochemical control rates with acceptable toxicity in low risk prostate cancer but efficacy data in unfavorable type prostate cancer is less convincing. CyberKnife-SBRT (CK-SBRT) can be used to escalate radiation dose delivery to the prostate while sparing normal tissue.

DETAILED DESCRIPTION:
The optimal radiation schedule for the curative treatment of prostate cancer remains unknown. Prostate cancer patients receiving radiation therapy are typically treated 5 days per week for 8-9 weeks. Recent data suggest that large radiation fraction sizes are radio-biologically favorable over lower fraction sizes in prostate cancer radiotherapy. The sensitivity of a tumor or normal tissue to fraction size of radiation can be approximated by the alpha-beta ratio. It has been suggested that the alpha/beta ratio for prostate cancer is actually as low as 1.5 implying that the current radiation therapy paradigm for prostate cancer treatment might be fundamentally flawed, as high fraction sizes would be expected to damage tumor more readily.

Typical prostate SBRT doses do not appear to have similar efficacy in higher risk prostate cancer suggesting even higher doses are required. Many techniques including dose escalated external beam radiation therapy (EBRT), proton therapy (PT) and brachytherapy have been employed to increase dose to the prostate. Data from the ASCEND-RT trial utilizing low dose rate brachytherapy boost showed a dramatic 21% improvement in biochemical control at 9 years favoring brachytherapy boost compared to conventional dose escalated EBRT radiation therapy. However, no corresponding benefit was identified in overall survival, incidence of bone metastases or prostate cancer specific mortality while a 3 fold increase in late urinary toxicity was noted.

SBRT is well tolerated with minimal acute and late side effects. In this protocol, CK-SBRT will be used to target the microscopic and gross disease in the prostate, seminal vesicles. An escalated dose of 40 Gy in 5 fractions will be delivered to the entire target volume while any nodules visible within the prostate gland on endorectal MRI will receive 50 Gy in 5 fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within 360 days of enrollment.
* Prostate Specific Antigen (PSA) documented within 90 days prior to registration.
* Clinical staging completed within 90 days of registration.
* No Nodal or Distant Metastases documented on CT or MRI of the pelvis and bone scan.
* Unfavorable Risk Prostate Carcinoma as Described is documented.
* No prior pelvic radiotherapy.
* No prior Trans-urethral resection of the prostate (TURP).
* Prostate volume < 100 cc
* American Urologic Association (AUA) score < 20
* No recent (within 5 years) or concurrent cancers other than non-melanoma skin cancers.
* Patient must have no medical or psychiatric illnesses that would interfere with treatment or follow-up.
* No implanted hardware adjacent to the prostate that would prohibit appropriate treatment planning and treatment delivery is allowed.
* Candidate for rectal spacer placement

Exclusion Criteria:

* Other cancer diagnosis other than non-melanoma skin cancer with 5 years
* Prostate size greater than 100cc
* AUA greater than 20
* Implanted hardware impacting imaging
* Metastatic prostate cancer
* Contraindication to hormone therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males with prostate cancer
Enrollment: 100 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2028-07-12 (Estimated)

PRIMARY OUTCOMES:
Bladder and Rectal Toxicity using NCI common toxicity criteria version 4.0 | 24 Months
  Genitourinary or Bowel Toxicity as a result of radiation therapy will be reported using

SECONDARY OUTCOMES:
Biochemical Disease Free Survival | 24 Months
  Time in months from completion of SBRT to biochemical failure
Duration of local control | 24 Months
  time in months from SBRT completion to local failure
Distant Failure | 24 Months
  time in months from SBRT completion to distant failure
Disease Free Survival | 24 Months
  time in months from the date that the patient is determined to be free of disease to the date of known disease recurrence for any measure of disease.
Disease Specific Survival | 24 Months
  time in months from completion of SBRT to death due to prostate cancer, other causes with active malignancy, or complications from treatment.
Overall Survival | 5 years
  ime in months from SBRT completion until death

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle Lanciano, MD, Study Chair — Philadelphia CyberKnife -Crozer Health; Rachelle Lanciano, MD, Principal Investigator — Philadelphia CyberKnife -Crozer Health
Locations (1):
- Philadelphia CyberKnife, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-06-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03822494/Prot_001.pdf